CLINICAL TRIAL: NCT06117189
Title: Turkish Validity and Reliability of Oral Health Impact on Daily Life Questionnaire in Endodontic Patients
Brief Title: Turkish Validity and Reliability of Oral Health Impact on Daily Life Questionnaire
Status: Completed | Type: Observational
Sponsor: Recep Tayyip Erdogan University (Other)
Responsible Party: Principal Investigator, Ahter Sanal Cikman, Assistant Professor, Recep Tayyip Erdogan University
Other Study IDs: 2023/118
Record Dates: First submitted 2023-10-20; First posted 2023-11-03 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-10

CONDITIONS: Oral Health Related Quality of Life
Keywords: oral health; quality of life
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult endodontic patients: Turkish version of Oral Health Impact on Daily Life questionnaire was applied to adult endodontic patients
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Oral Health Impact Daily Life questionnaire including 7 domains (eating, speaking, appearance, social, psychological, health, and finance) and 16 questions regarding perceived intensity

SUMMARY:
This study aimed to test Turkish validity and reliability of the Oral Health Impact on Daily Life Questionnaire (OHIDL) in adult endodontic patients.The questionnaire was translated and adapted into Turkish. Then, it was applied to two hundred twenty-two participants aged 18 years.

DETAILED DESCRIPTION:
This study aimed to test Turkish validity and reliability of the Oral Health Impact on Daily Life Questionnaire (OHIDL) in adult endodontic patients.

The questionnaire was translated and adapted into Turkish. Two hundred twenty-two participants aged 18 years and over without systemic disease were included. The reliability was examined by internal consistency and test-retest reliability. The construct and criterion validity were examined by evaluating the correlation of each question with the domains, the correlation of the domains with the global questions, and the correlation of Turkish-OHIDL with the Turkish version of the Oral Health Impact Scale (OHIP-14-TR). Statistical analysis was performed with SPSS 21.0 (IBM Corp, Armonk, NY, USA). P <0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and older who applied to the Department of Endodontics

Exclusion Criteria:

* Patients who did not speak Turkish,
* Patients having cognitive impairment,
* Patients having communication difficulties

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 years and older who applied to the Department of Endodontics
Sampling Method: Probability Sample
Enrollment: 222 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-07-15 (Actual)

PRIMARY OUTCOMES:
To asses Turkish validity and reliability of Oral Health Impact on Daily Life questionnaire | One month from the beginning of the study
  The reliability was examined by internal consistency and test-retest reliability. The construct and criterion validity were examined by evaluating the correlation of each question with the domains, the correlation of the domains with the global questions, and the correlation of Turkish-OHIDL with the Turkish version of the Oral Health Impact Scale (OHIP-14-TR).

CONTACTS AND LOCATIONS:
Overall Officials: Ahter Şanal Çıkman, Principal Investigator — Recep Tayyip Erdogan University
Locations (1):
- Recep Tayyip Erdogan University, Rize, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No